CLINICAL TRIAL: NCT01545518
Title: IVIG Treatment for Refractory Immune-Related Adult Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility criteria, unable for Phase 2 of study, & phase 1 was terminated.
Sponsor: Emory University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Charles M. Epstein, MD, Professsor of Neurology - Divsion of Epilepsy, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00052646; BT11-000312 (Other: Other)
Record Dates: First submitted 2011-11-30; First posted 2012-03-06 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Epilepsy, Cryptogenic; Epilepsy, Partial; Seizure Disorder; Autoimmune Diseases, Nervous System; Limbic Encephalitis
Keywords: Refractory epilepsy; Cryptogenic epilepsy; Autoimmune disorders; IVIG; Immunomodulatory therapy; Autoantibodies
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Autoimmune Diseases of the Nervous System; Limbic Encephalitis; Drug Resistant Epilepsy; Autoimmune Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental): IVIG
  Interventions: Drug: IVIG

INTERVENTIONS:
Drug: IVIG — IVIG 2 mg/kg in two divided doses with placebo crossover
  Other Names: IVIG manufactured by Baxter Healthcare Corporation

SUMMARY:
The purpose of the initial screening study is to find out if immune problems are an unrecognized cause of epilepsy in some patients. This study consists of a single blood sample, which will be tested for possible immune abnormalities. If enough patients are found who show immune abnormalities, those patients who are still having uncontrolled seizures will be invited to participate in a study of immune treatment with a compound called intravenous immunoglobulin (IVIG).

The study hypothesis is that a significant proportion of the young-onset, refractory, image-negative, partial-onset epilepsy population have an underlying autoimmune disorder, and many of these patients will respond to immune therapies, including IVIG.

At present, the importance of immune abnormalities in causing epilepsy, and the proper treatment when they are found, are both poorly understood. The investigators hope that this study will help us understand the cause of some cases that are difficult to treat.

DETAILED DESCRIPTION:
The study is divided into two phases:

Phase I: The investigators will screen for evidence of neuronal nuclear, cytoplasmic, and cell surface autoantibodies in our population of new onset refractory, imaging-negative young adult epilepsy patients. This part of the study involves obtaining a single blood sample, equal to about 2 teaspoons.

Phase 2: If a sufficient number of cases are identified, a double-blind crossover study of IVIG treatment will be performed in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uncontrolled epilepsy with at least two seizures a month for three consecutive months.
* Age 18 to 50.
* Clinical semiology or electroencephalogram (EEG) consistent with partial onset epilepsy.
* Refractory to an adequate trial of two or more main-line anti-epileptic drugs.
* Ability to keep a seizure diary.
* Normal brain magnetic resonance imaging (MRI) - 3 Tesla, seizure protocol; with the exception of hippocampal sclerosis

Exclusion Criteria:

* History of severe prematurity or neonatal distress, febrile seizures, moderate or sever traumatic brain injury, stroke, brain tumor, meningitis, encephalitis, neurocutaneous syndromes, or intracranial metal objects.
* Evidence of psychogenic epilepsy.
* History of convulsive status epilepticus.
* History of primary generalized epilepsy in a first degree relative.
* Known serious medical illness.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Epstein, M.D., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - The Emory Clinic, Inc., Atlanta, Georgia

REFERENCES:
- [Background] Alamowitch S, Graus F, Uchuya M, Rene R, Bescansa E, Delattre JY. Limbic encephalitis and small cell lung cancer. Clinical and immunological features. Brain. 1997 Jun;120 ( Pt 6):923-8. doi: 10.1093/brain/120.6.923. PMID 9217677
- [Background] Graus F, Keime-Guibert F, Rene R, Benyahia B, Ribalta T, Ascaso C, Escaramis G, Delattre JY. Anti-Hu-associated paraneoplastic encephalomyelitis: analysis of 200 patients. Brain. 2001 Jun;124(Pt 6):1138-48. doi: 10.1093/brain/124.6.1138. PMID 11353730
- [Background] Gultekin SH, Rosenfeld MR, Voltz R, Eichen J, Posner JB, Dalmau J. Paraneoplastic limbic encephalitis: neurological symptoms, immunological findings and tumour association in 50 patients. Brain. 2000 Jul;123 ( Pt 7):1481-94. doi: 10.1093/brain/123.7.1481. PMID 10869059
- [Background] Jacobs DA, Fung KM, Cook NM, Schalepfer WW, Goldberg HI, Stecker MM. Complex partial status epilepticus associated with anti-Hu paraneoplastic syndrome. J Neurol Sci. 2003 Sep 15;213(1-2):77-82. doi: 10.1016/s0022-510x(03)00130-8. PMID 12873758
- [Background] Lawn ND, Westmoreland BF, Kiely MJ, Lennon VA, Vernino S. Clinical, magnetic resonance imaging, and electroencephalographic findings in paraneoplastic limbic encephalitis. Mayo Clin Proc. 2003 Nov;78(11):1363-8. doi: 10.4065/78.11.1363. PMID 14601695
- [Background] Lucchinetti CF, Kimmel DW, Lennon VA. Paraneoplastic and oncologic profiles of patients seropositive for type 1 antineuronal nuclear autoantibodies. Neurology. 1998 Mar;50(3):652-7. doi: 10.1212/wnl.50.3.652. PMID 9521251
- [Background] McKeon A, Ahlskog JE, Britton JW, Lennon VA, Pittock SJ. Reversible extralimbic paraneoplastic encephalopathies with large abnormalities on magnetic resonance images. Arch Neurol. 2009 Feb;66(2):268-71. doi: 10.1001/archneurol.2008.556. PMID 19204167
- [Background] Nahab F, Heller A, Laroche SM. Focal cortical resection for complex partial status epilepticus due to a paraneoplastic encephalitis. Neurologist. 2008 Jan;14(1):56-9. doi: 10.1097/NRL.0b013e3181578952. PMID 18195661
- [Background] Pittock SJ, Kryzer TJ, Lennon VA. Paraneoplastic antibodies coexist and predict cancer, not neurological syndrome. Ann Neurol. 2004 Nov;56(5):715-9. doi: 10.1002/ana.20269. PMID 15468074
- [Background] Porta-Etessam J, Ruiz-Morales J, Millan JM, Ramos A, Martinez-Salio A, Berbel-Garcia A. Epilepsia partialis continua and frontal features as a debut of anti-Hu paraneoplastic encephalomyelitis with focal frontal encephalitis. Eur J Neurol. 2001 Jul;8(4):359-60. doi: 10.1046/j.1468-1331.2001.00213.x. No abstract available. PMID 11422434
- [Background] Shavit YB, Graus F, Probst A, Rene R, Steck AJ. Epilepsia partialis continua: a new manifestation of anti-Hu-associated paraneoplastic encephalomyelitis. Ann Neurol. 1999 Feb;45(2):255-8. doi: 10.1002/1531-8249(199902)45:23.0.co;2-n. PMID 9989630
- [Background] Thieben MJ, Lennon VA, Boeve BF, Aksamit AJ, Keegan M, Vernino S. Potentially reversible autoimmune limbic encephalitis with neuronal potassium channel antibody. Neurology. 2004 Apr 13;62(7):1177-82. doi: 10.1212/01.wnl.0000122648.19196.02. PMID 15079019
- [Background] Matarasso N, Bar-Shira A, Rozovski U, Rosner S, Orr-Urtreger A. Functional analysis of the Aurora Kinase A Ile31 allelic variant in human prostate. Neoplasia. 2007 Sep;9(9):707-15. doi: 10.1593/neo.07322. PMID 17898866
- [Background] Rudzinski LA, Pittock SJ, McKeon A, Lennon VA, Britton JW. Extratemporal EEG and MRI findings in ANNA-1 (anti-Hu) encephalitis. Epilepsy Res. 2011 Aug;95(3):255-62. doi: 10.1016/j.eplepsyres.2011.04.006. Epub 2011 May 12. PMID 21570256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled in a medical setting if eligible. Inclusion and exclusion criteria. A total of 20 patients with unexplained refractory epilepsy were screened and tested with a multiple panel for anti-neuronal antibodies.
Pre-assignment Details: In comparisons with our original futility criteria, it was apparent that the absence of more powerful findings, and the time it took to collect the ones we have, indicated the virtual impossibility of identifying enough patients with strong autoimmune findings to carry out Phase 2 of this study.
Period: Overall Study
Arm/Group | All Subjects
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 18-50 years of age, both male and female
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Immune Abnormalities
Description: neuronal nuclear, cytoplasmic, and cell surface autoantibodies
Time Frame: Screening visit
Population: No analysis occurred and study was terminated early due to subject numbers not eligible for the 2nd phase of the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- All Subjects: IVIG
  IVIG: IVIG 2 mg/kg in two divided doses with placebo crossover
  No AE's.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Study was terminated early. Subject eligibility for phase 2 not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No